CLINICAL TRIAL: NCT02100943
Title: Exhaled Nitric Oxide as a Biomarker of Gestational Obstructive Sleep Apnea and Persistence Postpartum
Brief Title: Exhaled NO as a Biomarker of Gestational OSA and Persistence Postpartum
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 00026736
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-06

CONDITIONS: Pregnancy; OSA
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA in Pregnancy: Pregnant women between 32 0/7 prior to 35 6/7 weeks gestation

SUMMARY:
This study will evaluate the presence or absence of Obstructive Sleep Apnea (OSA) in the third trimester of pregnancy and again postpartum.

DETAILED DESCRIPTION:
This is a prospective cohort study to evaluate the presence or absence of OSA in the third trimester of pregnancy and again postpartum. The investigators will use the Watch-PAT200® device as their accepted standard for diagnosis of obstructive sleep apnea.

When enrolled, women will be taught how to use the Watch-PAT200® via a company produced video that will be shown in the clinic and will be available via YouTube for review later if needed. They will also complete the Berlin Questionnaire. The patient will then use the Watch-PAT200® device overnight to evaluate for obstructive sleep apnea. This will be performed between 32-36 weeks gestation. Apnea-hypopnea indices (AHI) will be calculated and an AHI>5 will be considered diagnostic for OSA.

The next morning when the patient returns the Watch-PAT200® device they will exhale into the NIOX MINO® to assess their exhaled nitric oxide levels. This will be performed between 800-1000 am by one of the study personnel.

The patient will also wear the Watch-PAT200® device the first postpartum night. The entire process will be repeated between 6-8 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Female (> or equal 18 year of age)
* Pregnant between 32 0/7 prior to 35 6/7 weeks gestation
* Anticipated delivery at Forsyth Medical Center: Winston Salem, North Carolina

Exclusion Criteria:

* Illicit drug/Alcohol abuse
* Current treatment for obstructive sleep apnea
* Age <18 years
* Inability to speak/read English proficiently enough to give informed consent
* Usage of alpha blockers or short acting nitrates
* Permanent pacemaker
* Sustained non-sinus cardiac arrhythmias

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between 32 0/7 prior to 35 6/7 weeks gestation
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Difference in incidence of Obstructive Sleep Apnea (OSA) | 6-8 weeks postpartum
  The difference in incidence of OSA during the third trimester and postpartum. We assumed an incidence of 25% during the third trimester, reducing to 6% postpartum. Comparison will be made with McNemar's test on proportions at an α level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Street, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Forsyth Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Street LM, Aschenbrenner CA, Houle TT, Pinyan CW, Eisenach JC. Gestational Obstructive Sleep Apnea: Biomarker Screening Models and Lack of Postpartum Resolution. J Clin Sleep Med. 2018 Apr 15;14(4):549-555. doi: 10.5664/jcsm.7042. PMID 29609706